CLINICAL TRIAL: NCT06294405
Title: Development of a Database to Optimize the Results With Intraocular Lens Implants
Brief Title: Intraocular Lens Implant Registry Study
Status: Recruiting | Type: Observational
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Principal Investigator, Dr. med.Isabella Baur, Ophthalmologist, University Hospital Augsburg
Other Study IDs: 24-0010
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Intraocular Lens Complication; Intraocular Lens Rotation; Intraocular Lens Associated Postoperative Inflammation; Lens Opacities
MeSH Terms: conditions — Cataract | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intraocular lens Implantation — Intraocular lenses are implanted during cataract surgery to replace the human crystalline lens.

SUMMARY:
The goal of this registry study is to optimize the results with intraocular lens implants used in cataract surgery.

DETAILED DESCRIPTION:
A variety of intraocular lens implants are available for patients undergoing cataract surgery and new technologies are continuously being developed in this field.

In the planned monocentric retro- and prospective clinical study, a database to optimize outcomes with modern intraocular lens implants will be established to further improve anatomical and functional outcomes.

Patients treated with an intraocular lens implant will be included. The retrospective evaluation of data includes data routinely collected prior to study inclusion (preoperative, intraoperative, postoperative up to the 1st study visit). Prospectively, refraction, visual acuity, examination findings, intraocular pressure and complications are recorded 1-6 months postoperatively. Depending on the type of IOL, results of further non-invasive measurements are also recorded. Optional follow-up visits with the aforementioned examinations are possible up to 10 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Treatment with an intraocular lens implant 18 years of age or older Patient consent Full legal capacity

Exclusion Criteria:

Dementia Pregnancy Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who receive an intraocular lens are offered to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2029-02-14 (Estimated); Study Completion 2029-02-14 (Estimated)

PRIMARY OUTCOMES:
Functional results with different Intraocular lenses | 6 months
  Visual acuity with different intraocular lenses is determined.
Contrast sestivitiy with different Intraocular lenses | 6 months
  Contrast sensitivity with different intraocular lenses is determined.
Anatomical results. | 6 months
  Anatomical results with different intraocular lenses are determined.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Augsburg, Augsburg, Germany

IPD SHARING:
Plan to Share IPD: No